CLINICAL TRIAL: NCT01060462
Title: Efficacy According to Treatment Timing in Immunocompromised Patients Treated With Itraconazole Injection as an Empiric Antifungal Therapy
Brief Title: Observational Study Investigating the Response Rate of Itraconazole Injection in Treating Immunocompromised Patients
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015691
Record Dates: First submitted 2010-01-21; First posted 2010-02-02 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Hematological Malignancies; Neutropenia; Fever
Keywords: Defervescence rate; Defervescence timing; Itraconazole
MeSH Terms: conditions — Hematologic Neoplasms; Neutropenia; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 001: Pts. w/ neutropenic fever associated w/ hematologic malignancy Itraconazole 200 mg twice daily for 2 days for a total of 4 doses then 200 mg once daily for 12 days. After 14 days of IV administration itraconazole oral solution 200 mg twice daily should be continued for a total of 14 days until clinically significant resolution of neutropenia resolves
  Interventions: Drug: Pts. w/ neutropenic fever associated w/ hematologic malignancy

INTERVENTIONS:
Drug: Pts. w/ neutropenic fever associated w/ hematologic malignancy — Itraconazole 200 mg twice daily for 2 days for a total of 4 doses, then 200 mg once daily for 12 days. After 14 days of IV administration, itraconazole oral solution 200 mg twice daily should be continued for a total of 14 days until clinically significant resolution of neutropenia resolves

SUMMARY:
The purpose of this observational study is to examine the rate at which elevated body temperature (fever) is relieved by an itraconazole injection administrated to patients experiencing neutropenic fever . A neutropenic fever is an elevated body temperature that occurs at a time when the patient's white blood cell count is low. White blood cells aid the body's normal defenses against infection, so a fever during this period might make it difficult for the patient to fight infections.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, prospective and observational study enrolling approximately 440 patients. The primary objective of this study is to examine the fever response rate after itraconazole IV (directly into the vein) is administered for more than 3 days to patients with neutropenic fever based on investigator's discretion. Follow-up will be performed before and after administration and for 7 days after administration. Study population consists of the patients who visit a study center during the study period and are judged to have neutropenic fever associated with hematologic malignancy such as acute leukemia, hodgkin's lymphoma, non-hodgkin's lymphoma, myelodysplastic syndrome, and multiple myeloma. The decision to treat patients with itraconazole is as per physician discretion and doses are determined based upon approved labeling recommendations and physician discretion. The safety and efficacy of itraconazole administered beyond 29 days is not yet been established in the treatment of fever in neutropenic patients suspected of systemic fungal infection. Itraconazole 200 mg IV twice daily for 2 days, for a total of 4 doses, then 200 mg IV once daily for 12 days. After the administration for a total of 14 days, itraconazole oral solution 200 mg (20 ml) twice daily should be continued for a total of 14 days

ELIGIBILITY:
Inclusion Criteria:

* Patients with neutropenic fever who receive antineoplastic therapy or stem cell transplantation for acute leukemia, hodgkin's lymphoma, non-hodgkin's lymphoma, myelodysplastic syndrome, and multiple myeloma
* Patients who are recommended to receive itraconazole injection for treatment of acute leukemia, hodgkin's lymphoma, non-hodgkin's lymphoma, myelodysplastic syndrome, and multiple myeloma

Exclusion Criteria:

* Childbearing women who are pregnant or likely to be pregnant during the study period and male patients who are neither infertile nor willing to refrain from sexual relations but whose partner does not conduct an effective contraception (implant, injections, oral contraceptives, intrauterine device, etc.)
* Fever due to documented deep-seated fungal infection at the entry into the study (documented candidemia will be included)
* Significant hepatic and renal dysfunction
* Patients who, at the discretion of the investigator, are not eligible for the study participation based on warnings, precautions and contraindicated medications as listed in the package insert of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of the patients who visit a study center during the study period and are judged to have neutropenic fever associated with hematologic malignancy such as acute leukemia, hodgkin's lymphoma, non-hodgkin's lymphoma, myelodysplastic syndrome, and multiple myeloma
Sampling Method: Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Frequency rate at which fever is resolved and the time to fever resolution | after completion of the treatment of 3 to 14 days and after 7 days of follow up period

SECONDARY OUTCOMES:
Defervescence rate according to baseline result of Chest X-ray, CT (Computed tomography, a medical imaging method), Galactomannan test (diagnosis test for fungal infection) | after completion of 3 to 14 days of treatment and after 7 days of follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- [Derived] Kim SJ, Cheong JW, Min YH, Choi YJ, Lee DG, Lee JH, Yang DH, Lee SM, Kim SH, Kim YS, Kwak JY, Park J, Kim JY, Kim HG, Kim BS, Ryoo HM, Jang JH, Kim MK, Kang HJ, Cho IS, Mun YC, Jo DY, Kim HY, Park BB, Kim JS. Success rate and risk factors for failure of empirical antifungal therapy with itraconazole in patients with hematological malignancies: a multicenter, prospective, open-label, observational study in Korea. J Korean Med Sci. 2014 Jan;29(1):61-8. doi: 10.3346/jkms.2014.29.1.61. Epub 2013 Dec 26. PMID 24431907